CLINICAL TRIAL: NCT01517256
Title: Living Everyday Above-and-beyond Pain Research (LEAP): A Pilot Study Evaluating a Multidisciplinary Chronic Pain Group Therapy in a Primary Care Setting
Brief Title: A Pilot Study Evaluating a Multidisciplinary Chronic Pain Group Therapy in a Primary Care Setting
Acronym: LEAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DFM 09-595
Record Dates: First submitted 2012-01-16; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Primary care; Multidisciplinary group therapy; Embedded mixed-methods study
MeSH Terms: conditions — Chronic Pain

ARMS (2):
- Early Intervention Group (Experimental)
  Interventions: Behavioral: Living Everyday Above-and-beyond Pain (LEAP)
- Delayed Intervention Group (Placebo Comparator): Initially wait-listed and served as control group. But later participants underwent the experimental intervention.
  Interventions: Other: Wait-listed

INTERVENTIONS:
Behavioral: Living Everyday Above-and-beyond Pain (LEAP) — 8-week multidisciplinary group therapy aiming consisting of education about the nature of chronic pain, pacing and goal setting, mindfulness medication techniques, cognitive reflections on beliefs, impulses and obsessions, physical activation, and medication management.
  Arms: Early Intervention Group
Other: Wait-listed — Patients are wait-listed while awaiting participation to the LEAP program.
  Arms: Delayed Intervention Group

SUMMARY:
The investigators will evaluate the effectiveness of "Living Everyday Above-and-beyond Pain" (LEAP) program in the primary care setting. LEAP is a multidisciplinary chronic pain group therapy developed for the two clinic sites of McMaster Family Health Team: McMaster Family Practice and Stonechurch Family Health Centre. LEAP aims to improve patients'quality of life, interaction with the health care system and their health care utilization. This is a pilot study to evaluate mainly feasibility. The investigators will make use of both experimental and qualitative methods gather evidence of the programs success, strengths and weaknesses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* diagnosed with chronic pain

Exclusion Criteria:

* chronic pain related to cancer, pelvic pain or headache
* inability to speak or write in English
* patient is unable to attend and participate in group treatment sessions on their own
* substance use or mental health problems of a severity making group treatment participation impossible
* currently participating in another cognitive-behavioral pain management program
* patient is receiving palliative care or has been diagnosed with an illness expecting to cause death within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 8 months
  This will utilize the SF-36 QOL questionnaire.
Health care utilization | 8 months
  This will be based on a chart review to assess the number of consultations with their family physician and other clinicians (Nurse practitioners, registered nurse, dietitian, social worker).

SECONDARY OUTCOMES:
Qualitative process evaluation (Perceptions of participants regarding the intervention) | 16 months
  This outcome assesses the views of the participants regarding the strengths and weaknesses of the intervention. It will assess ways to improve the recruitment process and retention of participants in the group, satisfaction of the participants regarding the processes (group dynamics, time, format, contents, etc), perceptions of participants regarding the effectiveness of the program, and suggestion of participants regarding ways to improve the program.
Pain medication use | 8 months
  This will be based on a standardized questionnaire developed by the researchers and a chart review regarding request for early refill and increased dose of medications due to worsening of chronic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Family Practice Clinic, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Angeles RN, Guenter D, McCarthy L, Bauer M, Wolfson M, Chacon M, Bullock L. Group interprofessional chronic pain management in the primary care setting: a pilot study of feasibility and effectiveness in a family health team in Ontario. Pain Res Manag. 2013 Sep-Oct;18(5):237-42. doi: 10.1155/2013/491279. Epub 2013 Jul 19. PMID 23875181